CLINICAL TRIAL: NCT03583918
Title: A Prospective, Multi-center, Pilot Study to Evaluate the Efficacy of Micro-Excisional Skin Remodeling With Micro-Coring Device in the Treatment of Wrinkles and Skin Laxity of Face and Neck
Brief Title: Efficacy of Micro-excisional Skin Removal by Micro-coring Device in Treatment of Wrinkles and Laxity of Face and Neck
Acronym: MCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Optimization of MCD treatment; AIS 700-00022 (Other: Cytrellis Biosystems, Inc.)
Record Dates: First submitted 2017-08-16; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Laxity; Skin
Keywords: facial wrinkles; skin laxity; sagging skin
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Highthroughput Micro Coring Device (Experimental): Skin excision and removal with with Highthroughput Micro Coring device
  Interventions: Device: HighThroughput Micro Coring Device

INTERVENTIONS:
Device: HighThroughput Micro Coring Device — Assess Safety and Efficacy for skin treatments through micro-excisional skin removal with micro-coring device
  Other Names: skin micro-coring

SUMMARY:
This is a prospective, multi-center, pilot study evaluating effectiveness of micro-excisional skin remodeling by micro-coring skin in subjects meeting the Inclusion Criteria. Subjects will undergo bilateral treatment on the face and neck (upper and lower cheek, upper and lower lip, periocular and perioral areas, submandibular and middle neck, etc). The exact treatment area(s), choice of treatment density are left to the Investigator's discretion and subject's consent. Up to 3 treatments are allowed with a minimum of 30-day between the consecutive treatments.

DETAILED DESCRIPTION:
The study will enroll up to 50 subjects at 6-8 investigational sites. It will evaluating effectiveness of a micro-coring device for micro-excisional skin remodeling in subjects with moderate to severe wrinkles of face and neck who meet the Inclusion/Exclusion Criteria. The choice of treatment density is at the investigator's discretion with the subject's consent. Up to 3 treatments may be performed with a minimum of 30-day interval between the consecutive treatments. Subjects will undergo bilateral micro-coring of skin on the face and upper neck, including but not limited to upper and lower cheek, upper and lower lip, periocular and perioral areas, submandibular and upper neck. The exact area(s) of treatment are left to the Investigator's discretion and subject's consent.

The subjects will be evaluated at each visit and following data will be collected:

* The incidence and severity of systemic and local adverse events.
* Wrinkle severity score assessed using the Lemperle Wrinkle Severity Scale.
* Changes in skin laxity assessed by Laxity Scale.
* Canfield Image Analyses.
* Needle and/or punch biopsy (in some subjects).
* Overall aesthetic improvement using the following scales:
* Subject and PI Global Aesthetic Improvement Scale (GAIS)
* Subject Satisfaction Scale
* Rhytides and Laxity Scale
* Lower face assessment
* Investigator evaluation of device usability and functionality. Data Analysis: Analyses will be conducted per measurement tools listed. Statistical analysis will include but will not be limited to T tests, univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type 1, 2, or 3 as judged by the Investigator
* Two or more of the following: Facial wrinkles assessed using the Lemperle Wrinkle Assessment Scale (descriptive and pictorial)

  * Cheek fold lines >2
  * Upper lip lines >3
  * Nasolabial Folds >3
  * Marionette lines >3
  * Labiomental crease >3
  * Corner of the mouth lines >3
  * Periocular lines >3
* Able to provide written informed consent, understand and willing to comply with all study related directions from investigator and follow-up visits.

Exclusion Criteria:

* Lesions suspicious for any malignancy or the presence of actinic keratosis, melasma, vitiligo, cutaneous papules/nodules or active inflammatory lesions in the areas to be treated
* History of keloid formation or hypertrophic scarring
* History of trauma or surgery to the treatment areas in the past 6 months
* Scar present in the areas to be treated
* Silicone or synthetic material injections in the areas to be treated
* Injection of FDA-approved dermal fillers in the past two years
* Injection of fat in the past year
* History of treatment with dermabrasion, ablative laser, or radiofrequency in the past year
* History of treatment with non-ablative laser in the past 6 months
* History of treatment with botulinum toxin injections in the areas to be treated within the prior 6 months
* Active smokers (0.5 pack/day) or having quit within 3 months prior to treatment
* Active, chronic, or recurrent infection
* History of compromised immune system or currently being treated with immunosuppressive agents
* History of sensitivity to analgesic agents, Aquaphor®, topical or local anesthetics (e.g., lidocaine, benzocaine, procaine) or chlorhexidine, povidone-iodine or epinephrine
* Excessive sun exposure and use of tanning beds or tanning creams within 30 days prior to treatment
* Treatment with aspirin or other blood thinning agents within 14 days prior to treatment
* History or presence of any clinically significant bleeding disorder
* Co-morbid condition that in the Investigator's opinion could limit ability to participate in the study or to comply with follow-up requirements
* History of drug and/or alcohol abuse
* Any issue that, at the discretion of the Investigator, would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent
* Treatment with an investigational device or agent within 30 days before treatment or during the study period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Assess wrinkle reduction for moderate to severe wrinkles at 90 days post treatment based on the Lemperle Wrinkle Scale | 90-day post-treatment
  Assess wrinkle reduction in wrinkle severity score from the baseline assessed by Independent Reviewer(s) using the Lemperle Wrinkle Severity Scale. No wrinkles = 0; Just perceptible wrinkles = 1; Shallow wrinkles = 2; Moderately deep wrinkles = 3; Deep wrinkles, well-defined edges = 4; Very deep wrinkles, redundant fold = 5

SECONDARY OUTCOMES:
Assess skin laxity Improvement at 90 days post treatment | 90-day post-treatment
  Improvement in skin laxity score from the baseline assessed by Independent Reviewer using Laxity Scale and supplemented by the Canfield Image Analyses. Global Aesthetic Improvement Scale: 3 Very Much Improved; 2 Much Improved; 1 Improved; 0 No Change; - 1 Worse; - 2 Much Worse; -3 Very Much Worse.
Assess skin for new collagenases | 60, 90, 180-day post treatment
  Histological changes in treated skin when compared to untreated skin consistent with new collagenases

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Krantz, MBA, Study Director — Cytrellis Biosystems, Inc.
Locations (5):
- United States (5):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Miami Dermatology and Laser Institute, Miami, Florida
  - Laser and Skin Surgery Center of New York, New York, New York
  - The Practice of Brian S. Biesman, M.D, Nashville, Tennessee
  - Dr A Jay Burns Cosmetic Surgery, Dallas, Texas